CLINICAL TRIAL: NCT03202810
Title: Biomarker-driven Approach to Develop Population-wide Cost-effective Prevention Strategies for High-risk Oral Premalignancies
Brief Title: Innovative Approach to Triage Oral Precancer
Acronym: iTOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H11-02516
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Oral Cancer; Oral Premalignant Lesion
Keywords: optical imaging technology, loss of heterozygosity, prevention, miRNA, cost-effectiveness
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embeded biopsy specimens, blood samples for serum, plasma, and DNA; fresh frozen tissue of biopsy specimens; exfoliated cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral cancer is a major health problem worldwide, accounting for 274,000 new cases and 145,000 deaths annually. On average, half of the patients die within 5 years of an oral cancer diagnosis. Most troubling, however, is the lack of significant change in prognosis for this disease over the last 4 decades, even in developed nations. Even when successful, treatment of oral cancer can be devastating due to diminished quality of life and disfigurement. The key to controlling this disease is early identification of lesions that are at high risk of progression and provide effective treatment. The overall objective of the team is to integrate clinical, pathological, molecular, and imaging data to create a robust oral cancer risk model to predict the risk of progression of OPLs and to develop population-wide cost-effective prevention strategies for high-risk oral premalignancies. The project will involve 4 specific aims as described in detail below.

Aim 1. To use molecular data to stratify low-grade OPLs into high- and low-risk groups.

Aim 2. To evaluate the cost-effectiveness of various follow-up frequency that use LOH at chromosome 9p21 as a risk marker.

Aim 3: To evaluate the specificity and sensitivity of using imaging technologies as a tool for the decision of the high-grade or high-risk biopsy site.

Aim 4. To assess the clinical utility of a miRNA expression signature derived from serum collected from patients with oral cancer and OPLs.

DETAILED DESCRIPTION:
1. Patient accrual This study will be occurring at the Otolaryngology Clinic, Vancouver General Hospital. Three hundred and sixty volunteer subjects will be enrolled to participate in the study. Detailed steps of the study patient accrual are provided below.

   1. The establishment of referral pipelines for a true population-based OPL cohort in BC.

      In BC, the BC Oral Biopsy Service (OBS) and the Pathology Department at Vancouver General Hospital (VGH) receive biopsy and surgical specimens from the dental and medical communities, respectively. These centralized biopsy services offer a very rare opportunity to establish a population-based cohort of OPLs. The pathologists team will identify eligible patients through the pathology sign-out process and call the submitting physicians to notify the potential referral pipeline as an alternative management for these patients. Currently, a referral pipeline for severe dysplasia or more advanced oral malignancy using this model exists and has been established to refer surgical patients for the TFRI-funded COOLS trial (by Drs. Durham and Poh; H09-03090). This same system/pipeline will be used to identify eligible patients diagnosed with mild and/or moderate dysplasias identified from both medical and dental communities.
   2. Eligibility Subjects over the age of 19 attend the Dental or Otolaryngology clinic at the Vancouver General Hospital (Vancouver Acute) for assessment of oral lesions diagnosed with mild or moderate dysplasia; are willing to give the informed consent.
   3. Recruitment & informed consent procedures A letter of invitation regarding this study will be mailed to the potentially eligible patients a week before their appointment date along with the consent document. On the day of the clinical visit, the research assistant will explain the study to the eligible subject and acquire signed consent from the participants. 400 subjects will be recruited. These patients will be monitored once every six months (the current standard of care). When clinically warranted due to signs of disease progression or at the 2-year follow-up mark, two 5-mm punch biopsies will be performed on lesion areas with different severity (as determined by imaging technologies). Two-year comparative biopsy at a stable lesion is current standard of care.
2. Study procedures The study is a longitudinal study following the follow-up schedule of the current standard of care for such lesions, i.e., once per 6 months and comparative biopsy once per 2-3 years. The important time points are initial visit (baseline), at the end of second, 5th and 8th year of follow up visits. However, the time of biopsy is solely based on the clinical judgment of the clinicians, i.e., signs of disease progression.

   1. Clinical data collection After the subject has consented, they will be asked to complete a set of questionnaires for the collection of demographics and risk factor information. The subject will be assigned a study ID and no unique identifier will be linked to the data collected. A separate file will be used to link the study ID and patient identifiers. This is important to facilitate patient management and capture the outcome information. This file with patients' unique identifier will be kept in the pass-word protected file in the BC Cancer Research Centre (BCCRC) computer in a locked office in the BCCCRC and only PIs can access the file. The health status and HAI questionnaire is not for diagnostic purposes. Should the clinicians believe there is depression or anxiety present in the participant (clinicians' clinical judgment), the study clinicians in charge of this specific participant will communicate with patient's family doctor and refer the participant to a proper source for further evaluation and management.
   2. Data collection using study device

      * The clinicians will examine the patients using WL, VELScope VX for FV (previously approved, R05-0116), OCT (previously approved, H09-01955), and a hand-held confocal microscope (H11-00011).
      * OCT imaging: After identifying the abnormal areas for biopsy using WL and FV examination, the clinician will place a fiber-optic probe of the OCT on the oral mucosal areas of interest. The site for placement of the probe will be determined by PIs (Otolaryngology-head and neck surgeons (SD/DA) and/or Oral Medicine/Oral Pathology Specialist (Ng/Poh)). The images will be recorded by the machine for later analysis.
      * Confocal microscope imaging: After OCT imaging, the clinician will apply 0.05% Acriflavine Hydrochloride solution topically on the oral mucosal areas of interest for 30 seconds prior to imaging. The clinician will place a hand-held confocal microscope on the mucosal surface to record the observation for later analysis.
      * All necessary efforts will be taken to reduce any mild discomfort that could be associated with the probe placement inside the oral cavity of a subject. The OCT probe or the confocal microscope will be covered by a plastic barrier and disinfected by standard methods used for oral cavity instruments before and after subject usage. The device examination will take no more than 15 minutes in addition to the subject's appointment time for their routine visits. The maximum intensity of tissue illumination for each measurement will be less than the Threshold Limit Value (TLV) established by the American Conference of Governmental Industrial Hygienists (ACGIH)11 for exposure to broadband light.
      * The information obtained from polarized reflectance measurements will be compared with the histology and quantitative pathology (nuclear phenotype score) of the tissue sections from the lesion. The collected spectra data from normal looking areas from adjacent normal looking mucosa and contralateral mucosa will be used to determine patient to patient variation in the polarized reflectance of oral mucosa.
   3. Exfoliative brushing sample collection (previously approved, R05-0116) An Innovatec cytology brush (Arcona Inc) is used to collect exfoliated cells from the oral lesion. These brushings are transferred into PreservCyt® Solution (Cytyc Corp.) and keep in 4ºC fridge.
   4. Blood sample collection In total, 12 ml (3/4 of a tablespoon) of blood sample will be collected in 1 SST and 1 EDTA vacutainers in the clinic by trained research personnel. The blood sample will be processed and serum, plasma and puffy coat samples will be aliquot and frozen in -80ºC for future analysis. The DNA samples in the puffy coat will be extracted and used as the normal control sample for the loss of heterozygosity (LOH) analysis. A separate consent will be used for this purpose. We anticipate that all aliquots of serum, plasma and puffy coat will be used up. Any remaining tissue will not be discarded or sold, but will be stored in a locked freezer room at the BC Cancer Agency for a period of up to fifteen years so that results of this study can be confirmed.
   5. Frozen tissue collection In the event of biopsy, tissue will be bisected. Half of the sample will be fixed in the formalin solution and sent to the pathology laboratory for analysis as a normal part of medical diagnosis procedure. Part of this tissue will be kept and used only after the diagnosis has been made. At no time will tissue be removed solely for the purpose of research. The donated tissue will be given a code for identification by the project leader, and will be kept in secure freezers at the BC Cancer Agency until genetic material (DNA and RNA) has been extracted for analysis. A separate consent will be used for this purpose. We anticipate that all donated tissue will be used up. Any remaining tissue will not be discarded or sold, but will be stored in a locked freezer room at the BC Cancer Agency for a period of up to fifteen years so that results of this study can be confirmed.
   6. Tissue microdissection and DNA extraction. The formalin-fixed, paraffin-embedded tissue blocks of the initial biopsy and biopsy from the follow-up visit will be obtained from the Department of Anatomical Pathology, the Vancouver General Hospital. at the time of clinical change or at 24 months follow-up visit will be requested for processing. Ten 10-µm thick sections for DNA sample, 2 4-µm unstained tissue sections for quantitative histological analysis. Areas of dysplasia on the thick sections will be identified and microdissected. The DNA sample from the epithelium will be extracted and used for the LOH analysis.

ELIGIBILITY:
Inclusion Criteria:

* Is age 19 or older
* Have an abnormal lesion in the mouth.
* able to give informed consent to participate

Exclusion Criteria:

* less than 19 years old

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathology-proven oral precancers, i.e., verrucous hyperplasia, mild dysplasia, moderate dsyplasia are willing to give informed consent for the study.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2011-11-15 (Actual); Primary Completion 2021-11-14 (Estimated); Study Completion 2022-11-14 (Estimated)

PRIMARY OUTCOMES:
Cancer progression | 10 years
  the lesion progresses into high-grade preinvasive lesion or cancer

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Poh, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided